CLINICAL TRIAL: NCT06224907
Title: GENEr8-JPN: A Phase 3 Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of BMN 270, an Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Japanese Hemophilia A Patients With Residual FVIII Levels ≤ 1 IU/dL Receiving Prophylactic FVIII Infusions
Brief Title: Phase 3 Study for Efficacy and Safety Outcomes Data in Japanese Patients With Severe Hemophilia A
Acronym: GENEr8-JPN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 270-304
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia A
Keywords: Gene Therapy; Clotting Disorders; Blood Disorder; Blood Coagulation Disorders; Inherited Blood Coagulation disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases; Inborn; Factor VIII; Coagulants
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders; Hematologic Diseases; Blood Coagulation Disorders; Blood Coagulation Disorders, Inherited; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — Valoctocogene Roxaparvovec

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valoctocogene roxaparvovec (Experimental): Single administration of valoctocogene roxaparvovec at a dose of 6E13 vg/kg
  Interventions: Biological: Valoctocogene roxaparvovec

INTERVENTIONS:
Biological: Valoctocogene roxaparvovec — Adeno-Associated Virus Vector-Mediated Gene Transfer of Human Factor VIII in Severe Hemophilia A
  Other Names: BMN 270, ROCTAVIAN

SUMMARY:
This Phase III clinical study will evaluate the safety and effectiveness of valoctocogene roxaparvovec in Japanese patients with severe hemophilia A.

DETAILED DESCRIPTION:
This is a Phase 3, single-arm, open-label study in Japanese hemophilia A (HA) participants with endogenous coagulation factor VIII (FVIII) activity levels <1 IU/dL treated continuously with prophylactic exogenous FVIII for a minimum of 1 year prior to enrollment. Participants will be enrolled at approximately 10 sites in Japan. Participants must have high-quality, well-documented historical data available concerning previous bleeding episodes and exogenous FVIII usage over the previous 12 months in order to be eligible to enroll in the study. Approximately 6 Japanese adult participants with severe HA will receive a 6E13 vg/kg dose of BMN 270 as a single intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males ≥18 years of age with HA and endogenous FVIII activity levels <1 IU/dL as evidenced by medical history, at the time of signing the informed consent
* Must have been on prophylactic FVIII replacement therapy for at least 12 months prior to study entry. High-quality, well-documented historical data concerning bleeding episodes and FVIII usage over the previous 12 months must be available.
* Treated/exposed to FVIII concentrates for a minimum of 150 exposure days.
* Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any study-related procedures.
* No previous documented history of a detectable FVIII inhibitor, and results from a Bethesda assay or Bethesda assay with Nijmegen modification of less than 0.6 Bethesda Units (BU) or less than 1.0 BU for laboratories with a historical lower sensitivity cutoff for inhibitor detection of 1.0 BU on 2 consecutive occasions at least 1 week apart within the past 12 months (at least 1 of which should be tested at the central laboratory).
* Sexually active participants must agree to use an acceptable method of effective contraception
* Willing to abstain from alcohol consumption for at least the first 52 weeks following BMN 270 infusion.

Exclusion Criteria:

* Detectable pre-existing antibodies to the AAV5 capsid.
* Any evidence of active infection or any immunosuppressive disorder, except for human immunodeficiency virus (HIV) infection. HIV-positive participants who meet all other eligibility criteria may be included.
* Significant liver dysfunction
* Most recent, prior FibroScan or liver biopsy showing significant fibrosis
* Evidence of any bleeding disorder not related to HA.
* Platelet count of <100E9/L.
* Creatinine ≥1.5 mg/dL.
* Liver cirrhosis of any etiology as assessed by liver ultrasound.
* Chronic or active hepatitis B
* Active hepatitis C
* Active malignancy, except non-melanoma skin cancer
* History of hepatic malignancy
* History of arterial or venous thromboembolic events
* Known inherited or acquired thrombophilia, including conditions associated with increased thromboembolic risk, such as atrial fibrillation
* Treatment with any investigational product (IP) within 30 days or 5 half-lives of the IP prior to the Screening period.
* Any condition that, in the opinion of the investigator or sponsor would prevent the participant from fully complying with the requirements of the study
* Prior treatment with any vector or gene transfer agent.
* Major surgery planned in the 52-week period following the infusion with BMN 270.
* Use of systemic immunosuppressive agents, not including corticosteroids, or live vaccines within 30 days before the BMN 270 infusion.
* Concurrent enrollment in another clinical study unless it is an observational (non-interventional) clinical study that does not interfere with the requirements of the current protocol or have the potential to impact the evaluation of efficacy and safety of BMN 270 and with prior consultation with the medical monitor.
* Known allergy or hypersensitivity to BMN 270 IP formulation.
* Unwilling to receive blood or blood products for treatment of an AE and/or a bleeding episode.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in the human coagulation factor VIII (hFVIII) activity, as measured by chromogenic substrate assay, during Weeks 49 to 52 post BMN 270 infusion from Baseline. | 52 Weeks
  The change from baseline in FVIII activity, as measured by chromogenic substrate assay, during Weeks 49 to 52 post-BMN 270 infusion.
  Each subject's FVIII activity level during Week 49 to 52 is defined as the median of the values obtained during week 49-52 with the analysis window defined.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis. The baseline value is imputed as 1 IU/dL for each subject.

SECONDARY OUTCOMES:
Change in the annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy in the efficacy evaluation period (EEP) ("Post FVIII Prophylaxis to Last Visit") from the Baseline utilization of exogenous FVIII replacement therapy. | Baseline to at least Week 52
  The change from baseline in the annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy in the EEP period .
  The annualized utilization (IU/kg/year) of exogenous FVIII replacement therapy is defined as Sum of FVIII use (IU/kg) during calculation period/Total number of days during the calculation period ×365.25.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis. EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or 3 days post the end of FVIII prophylaxis ), whichever is later, to last visit by the data cut-off for the 1-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Change in the annualized bleeding rate (i.e., number of bleeding episodes per year) requiring exogenous FVIII replacement treatment therapy in the efficacy evaluation period ("Post FVIII Prophylaxis to Last Visit") from Baseline. | Baseline to at least Week 52
  ABR for treated bleeds=Number of bleeding episodes for treated bleeds during the calculation period/total number of days during the calculation period * 365.25 Bleeds that were treated with FVIII replacement therapy (recorded as "treatment for bleed") within 72 hours and were not associated with surgery or a procedure were included.
  Baseline: prior to BMN 270 infusion while receiving FVIII prophylaxis. EEP: From Week 5 post-BMN 270 infusion (Study Day 33) or 3 days post the end of FVIII prophylaxis , whichever is later, to last visit by the data cut-off for the 1-year analysis, hereafter referred to as "Post FVIII Prophylaxis to Last Visit").
Change from Baseline in Hemophilia-Specific Health-Related Quality of Life Questionnaire for Adults (Haemo-QoL-A) total score, physical functioning, role functioning, and consequences of bleeding domain scores at Week 52 of study post-BMN 270 infusion | Baseline to Week 52
  The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 52 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks).
  The Haemo-Qol-A physical functioning domain score is an average of each item value within a domain. The range of domain scores is 0 to 5; higher scores mean better HRQoL or less impairment for the domain. The physical functioning domain score is transformed to a 0 (minimum) to 100 (maximum) scale with higher scores indicating a better or less impaired haemophilia-related physical functioning
Change from Baseline in the Haemo-QoL-A worry, emotional impact, and treatment concern domain scores at Week 52 of the study post-BMN 270 infusion. | Baseline to Week 52
  The change from baseline (assuming no treatment for severe hemophilia A) in Haemo-Qol-A score, at week 52 post-BMN 270 infusion. The Haemo-Qol-A questionnaire is a fit for purpose hemophilia-specific health related quality of life (HRQoL) questionnaire for adults consisting of 41 items covering six domains (Physical Functioning, Role Functioning, Worry, Consequences of Bleeding, Emotional Impact and Treatment Concerns).The Haemo-Qol-A items are answered on a 6-point Likert scale ranging from 0 (none of the time) to 5 (all of the time).The recall period for the Haemo-Qol-A is one month (4-weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- Japan (4):
  - Asahikawa Medical University Hospital, Hokkaido, Asahikawa
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Nagoya University Hospital, Aichi, Nagoya
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku